CLINICAL TRIAL: NCT05143684
Title: Impact of Maternal Lateral Tilt on Cardiac Output During Caesarean Section Under Spinal Anaesthesia: A Prospective Observational Study
Brief Title: Maternal Lateral Tilt and Cardiac Output in Caesarean Section
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SONNINO CHIARA, Registered Anesthesiologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: LUD-CS
Record Dates: First submitted 2021-10-24; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Hypotension Drug-Induced
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Left Lateral Uterine Displacement — a wooden wedge wrapped with cotton, to make it comfortable, and medical sheets with a measured angle of 15° under the right flank of the laying down patient

SUMMARY:
Background: Left uterine displacement (LUD) has been questioned as an effective strategy to prevent aortocaval compression after spinal anesthesia (SA) for cesarean delivery (CD). The investigators tested if LUD has a significant impact on cardiac output (CO) in patients undergoing CD under SA during continuous non-invasive hemodynamic monitoring.

Methods: Forty-six patients were included in the final analysis. The investigators considered 4 timepoints of 5 minutes each: T1=baseline with LUD; T2=baseline without LUD; T3=after SA with LUD; T4=after SA without LUD. LUD was then repositioned for CD. Primary outcome was to test if CO decreased from T3 to T4. We also compared CO between T1 and T2 and other hemodynamic variables: mean, systolic and diastolic blood pressure (respectively MAP, SAP and DAP), heart rate (HR), stroke volume (SV), stroke volume variation (SVV), pulse pressure variation (PPV), contractility (dP/dt), dynamic arterial elastance (Eadyn) at the different timepoints. Data on fetal Apgar scores and umbilical arterial and venous pH were collecte

DETAILED DESCRIPTION:
The primary outcome was to test if CO decreases significantly after LUD removal in patients under SA for CD. This is a prospective observational study.

Data were gathered from pregnant patients who, in addition to standard monitoring, underwent perioperative non-invasive hemodynamic monitoring by ClearSight system on the Edwards Lifesciences HemoSphere platform (Edwards Lifesciences, Irvine, CA).

The parameters were recorded at 20 seconds-intervals. The investigators considered 4 timepoints. T1 were the baseline values recorded for 5 minutes, after initial stabilization of parameters, with the patient laying down on the operating table with LUD. At T2, LUD was removed and we considered for the analysis hemodynamic data of the subsequent 5 minutes. The investigators indicated as T3 the 5 minutes following SA with a satisfactory sensory block and as T4 the subsequent 5 minutes following LUD removal. Figure 1 summarizes the timepoints of our analysis. LUD was accomplished by positioning a wooden wedge wrapped with cotton, to make it comfortable, and medical sheets with a measured angle of 15° under the right flank of the laying down patient. In all patients, after T4 the 15° wooden wedge was positioned again and surgery was performed with LUD.

Anesthesia was standard spinal procedure, fluid management was left to the attending anesthesiologist.

The attending anesthesiologist was blinded to the advanced hemodynamic parameters from the ClearSight system except for the continuous BP values. The investigators defined hypotension as an absolute value of MAP < 65 mmHg. This value was considered as trigger for the attending anesthesiologist for the administration of norepinephrine 5 mcg. Norepinephrine boluses were repeated to reach a MAP>65mmHg. Bradycardia was defined as a heart rate of < 60 bpm. Atropine 0.5 mg was administered for the treatment of bradycardia combined with hypotension, or for an absolute value of heart rate < 45 bpm. After delivery, Oxytocin was administered to facilitate the uterine contraction.

We also evaluated the impact of maternal blood pressure and CO on fetal outcome collecting neonatal Apgar scores at 1 and 5 minutes after birth, and umbilical cord arterial and venous pH.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients at term (36th to 40th week of gestation) scheduled for elective caesarean section under spinal anesthesia.

Exclusion Criteria:

* age <18 years
* American Society of Anesthesiologists score >3
* cardiac arrhythmias or aortic regurgitation
* pregnancy-induced hypertension
* pre-eclampsia
* body mass index (BMI) > 35 kg/m2
* foetal complications
* coagulation disorders or contraindication to neuraxial block
* emergency surgery
* preoperative infection
* patient's refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study only involves female pregnant patients at term scheduled for elective caesarean section.
Study Population: Patients scheduled for elective caesarean section under spinal anesthesia at IRCCS Fondazione Policlinico Universitario Agostino Gemelli
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiac Output (l/min) measured by non-invasive hemodynamic monitoring | at 5 minutes from left lateral uterine tilt removal under spinal anesthesia
  Does cardiac output decrease significantly after left lateral uterine displacement removal in patients under spinal anesthesia for caesarean delivery?

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano A Draisci, MD, Study Director — IRCCS Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sonnino C, Frassanito L, Piersanti A, Giuri PP, Zanfini BA, Catarci S, Draisci G. Impact of maternal lateral tilt on cardiac output during caesarean section under spinal anaesthesia: a prospective observational study. BMC Anesthesiol. 2022 Apr 11;22(1):103. doi: 10.1186/s12871-022-01640-6. PMID 35410115